CLINICAL TRIAL: NCT02885727
Title: Phase II Trial of in Situ Tumor Vaccination Using Durvalumab and "Booster" Radiation Therapy in Patients With Metastatic Adenocarcinoma of the Pancreas Who Have Progressed Through First-line Chemotherapy
Brief Title: Durvalumab Plus "Booster" RT for Metastatic Adenocarcinoma Pancreas Cancer Post Chemotherapy (GCC 1598)
Acronym: Panc-Durval+RT
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding issues caused the study to not be opened the at local IRB
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Department of Radiation Oncology, Principal Investigator, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00070528
Record Dates: First submitted 2016-08-19; First posted 2016-08-31 (Estimated); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Metastatic Pancreas Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — durvalumab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Durvalumab + Radiation therapy (Experimental): Durvalumab (MEDI4736) 750 mg (or 10mg/kg if the patient weighs <30 kg) IV Q2W over 1 hour for all patients + Radiation therapy
  * First lesion to receive 25 Gy / 5 daily consecutive fractions of 5 Gy
  * Second lesion to receive15 Gy / 5 daily consecutive fractions
  Interventions: Drug: Durvalumab; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Durvalumab — Evaluate if the combination of RT and durvalumab can improve median PFS compared to chemotherapy historical control data in metastatic pancreas cancer patients who have progressed through first-line chemotherapy
  Other Names: (MEDI4736)
Radiation: Radiation Therapy — The primary intent of RT in this study is to augment a pancreatic cancer-specific immune response when given with durvalumab.

SUMMARY:
Research Hypothesis: The combination of ionizing radiation and immunotherapy (durvalumab) is well tolerated and stimulates a clinically significant pancreas-cancer specific immune response.

The primary objective will be to evaluate whether the combination of RT and durvalumab can improve median PFS compared to chemotherapy historical control data in metastatic pancreas cancer patients who have progressed through first-line chemotherapy.

The primary intent of RT in this study is to augment a pancreatic cancer-specific immune response when given with durvalumab.

DETAILED DESCRIPTION:
This clinical trial will use the combination of ionizing radiation and immunotherapy durvalumab (MEDI4736). It is the investigators hypothesis that this combination of ionizing radiation and immunotherapy is well tolerated and stimulates a clinically significant pancreas-cancer specific immune response. This trial's primary objective will be to evaluate whether the combination of RT and durvalumab can improve median PFS compared to chemotherapy historical control data in metastatic pancreas cancer patients who have progressed through first-line chemotherapy. The study population includes the metastatic pancreatic adenocarcinoma patients who have progressed through first-line chemotherapy. The number of subjects proposed to complete this study is 55.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and any locally-required authorization (e.g., HIPAA in the USA, EU Data Privacy Directive in the EU) obtained from the subject prior to performing any protocol-related procedures, including screening evaluations
2. Age > 18 years at time of study entry.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Life expectancy of ≥12 weeks as estimated by the investigator.
5. Biopsy-proven metastatic pancreatic adenocarcinoma with progression through standard first-line chemotherapy. Chemotherapy given as part of prior chemoradiation in the setting of non-metastatic pancreatic cancer does not count as a line of therapy.
6. ≥2 radiographically distinct and measurable pancreatic cancer lesions (primary and/or metastatic lesions) by RECIST 1.1 criteria separated by ≥5 cm
7. No lesion that would receive RT >7 cm in greatest dimension.
8. Subjects must consent to all study procedures described in the protocol including radiographic evaluation and repeated blood draws.
9. Adequate normal organ and marrow function as defined below:

   * Hemoglobin ≥ 9.0 g/dL
   * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L (> 1500 per mm3)
   * Platelet count ≥ 100 x 109/L (>100,000 per mm3)
   * Serum bilirubin ≤ 1.5 x institutional upper limit of normal (ULN). This will not apply to subjects with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.
   * AST (SGOT)/ALT (SGPT) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be ≤ 5x ULN
   * Serum creatinine CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance:

   Males:

   Creatinine CL (mL/min) = Weight (kg) x (140 - Age) / . 72 x serum creatinine (mg/dL)

   Females:

   Creatinine CL (mL/min) = Weight (kg) x (140 - Age) x 0.85 / 72 x serum creatinine (mg/dL)
10. Female subjects must either be of non-reproductive potential, not breast-feeding or must have a negative urine or serum pregnancy test within 28 days of study treatment, confirmed prior to treatment on day 1. Male or female patients of reproductive potential need to employ two highly effective and acceptable forms of contraception throughout their participation in the study and for 90 days after last dose of study drug.
11. Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

1. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site)
2. Previous enrollment in the present study
3. Any previous treatment with a PD1 or PD-L1 inhibitor, including durvalumab
4. Prior RT to any lesion that would receive RT on this protocol.
5. Prior RT that could lead to an unacceptably high risk of clinically significant normal tissue injury due to high cumulative normal tissue dose as determined by the investigator.
6. Subjects who have received second-line or later chemotherapy for metastatic pancreatic cancer (prior chemotherapy received in the non-metastatic setting does not count).
7. History of another primary malignancy except for:

   * Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of study drug and of low potential risk for recurrence
   * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
   * Adequately treated carcinoma in situ without evidence of disease e.g., cervical cancer in situ
8. Receipt of the last dose of anti-cancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies, other investigational agent) ≤14 days prior to the first dose of study drug.
9. Mean QT interval corrected for heart rate (QTc) ≥470 ms calculated from 3 electrocardiograms (ECGs) using Fridericia's Correction
10. Current or prior use of immunosuppressive medication within 28 days before the first dose of durvalumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid
11. Any unresolved toxicity (>grade 2, CTCAE version 4.03) from previous anti-cancer therapy. Subjects with irreversible toxicity that is not reasonably expected to be exacerbated by the investigational product may be included (e.g., hearing loss, peripherally neuropathy.
12. Any prior Grade ≥3 immune-related adverse event (irAE) while receiving any previous immunotherapy agent, or any unresolved irAE >Grade 1
13. Active or prior documented autoimmune disease within the past 2 years NOTE: Subjects with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded.
14. Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis)
15. History of primary immunodeficiency
16. History of allogeneic organ transplant
17. History of liver cirrhosis and Child-Pugh class B or C
18. History of hypersensitivity to durvalumab or any excipient
19. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses, any subject known to have evidence of acute or chronic hepatitis B, hepatitis C or human immunodeficiency virus (HIV), or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent
20. Known history of previous clinical diagnosis of tuberculosis
21. History of leptomeningeal carcinomatosis
22. Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving durvalumab
23. Female subjects who are pregnant, breast-feeding or male or female patients of reproductive potential who are not employing an effective method of birth control
24. Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results
25. Symptomatic or uncontrolled brain metastases requiring concurrent treatment, inclusive of but not limited to surgery, radiation and/or corticosteroids.
26. Subjects with uncontrolled seizures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-07 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Improvement in median Progression Free Survival using the combination of RT and durvalumab. | 6 years
  The primary objective will be to evaluate whether the combination of RT and durvalumab improves median PFS compared to historical control in metastatic pancreas cancer patients who have progressed through first-line chemotherapy. PFS is defined as the time from the date of durvalumab initiation to the date of pancreatic cancer progression or death, whichever occurs first. This is a clinically relevant and appropriate endpoint for a phase II trial and since there are no prior studies using immune checkpoint blockade with concurrent RT for metastatic pancreatic cancer will allow for historical comparison to PFS using second-line chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Shahed N Badiyan, MD, Principal Investigator — University of Maryland, Baltimore

IPD SHARING:
Plan to Share IPD: No